CLINICAL TRIAL: NCT05071222
Title: A Phase 1/2 Open Label Non Randomized Study, Multicentric, Single Arm Evaluating the Safety and Efficacy of Gene Therapy of the Severe Combined Immunodeficiency (SCID) Caused by Mutations in the Human DCLRE1C Gene (Artemis) by Transplantation of a Single Dose of Autologous CD34+ Cells Transduced ex Vivo With the G2ARTE Lentiviral Vector Expressing the DCLRE1C cDNA
Brief Title: Safety and Efficacy Study of Transplantation of Autologous CD34+ Cells Transduced With the G2ARTE Lentiviral Vector Expressing the DCLRE1C cDNA in Artemis (DCLRE1C) Deficient Severe Combined Immunodeficiency Patients (ARTEGENE)
Acronym: ARTEGENE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20180302; 2019-003555-11 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-10-08 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Artemis (DCLRE1C ) Deficient Severe Combined Immunodeficiency
Keywords: Artemis deficient Severe Combined Immunodeficiency; Severe Combined Immunodeficiency; Gene therapy; Allogeneic hematopoietic stem cells transplantation
MeSH Terms: conditions — Severe combined immunodeficiency with sensitivity to ionizing radiation; Xeroderma Pigmentosum, Complementation Group F; Severe Combined Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARTEGENE drug product (Experimental): Autologous purified CD34+ cells transduced with a self-inactivated lentiviral vector, expressing the DCLRE1C gene (alias Artemis)
  Interventions: Genetic: ARTEGENE drug product

INTERVENTIONS:
Genetic: ARTEGENE drug product — Each patient will receive a single intravenous infusion of ARTEGENE drug product at D0.

SUMMARY:
The purpose of this study is to evaluate the Safety and Efficacy of Gene Therapy of the severe combined immunodeficiency (SCID) caused by mutations in the human DCLRE1C gene (Artemis) by transplantation of a single dose of autologous CD34+ cells transduced ex vivo with the G2ARTE lentiviral vector expressing the DCLRE1C cDNA.

ELIGIBILITY:
Inclusion Criteria:

* Patient to 47 months
* SCID patients with confirmed biallelic mutations in the Artemis (DCLRE1C) gene even in the case of leaky forms characterised by a residual activity
* Absence of an HLA genoidentical donor or without rapidly available HLA-compatible unrelated donor (within six weeks of diagnosis)
* The patient can be treated by gene therapy without delay in case of active life threatening infections compromising the short-term prognosis and for which the delay in finding a phenoidentical donor is incompatible with the patient's condition of health. Active life threatening infections are defined as: viral respiratory infection, CMV infection, adenovirus infection, disseminated BCGitis or other infections grade ≥ 4 according to CTCAE scale
* Beneficiary of a social security scheme
* Parental, guardian's patient signed informed consent.

Exclusion Criteria

* Unwillingness to return for follow-up during the first 2 years study and the long term follow-up
* HIV-1 or 2 or HTLV1 infections
* Hypersensitivity to G-CSF, busulfan or Fludarabine
* Unable to tolerate general anesthesia and/or marrow harvest or peripheral blood stem cell collection (apheresis) or insertion of central venous catheter.

Max Age: 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2041-07-19 (Estimated); Study Completion 2041-07-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of transplant related mortality | Up to 100 days post treatment
Incidence of transplant related mortality | At 6 months post treatment
Transgene copy number on peripheral blood mononuclear cells (PBMCs) | Up to 15 years post treatment
  by qPCR
Transgene copy number on sorted cell populations | Up to 15 years post treatment
  Determined on sorted cell populations CD15+,CD14+, CD19+, CD56+ and CD3+ T lymphocytes by qPCR
Detection of replication-competent lentivirus (RCL) | 3 months post treatment
Absence of any severe adverse events due to insertional mutagenesis | Up to 15 years post treatment
Change in Artemis mRNA levels | At Day 0, 12 months and 24 months post treatment
  by RT-qPCR performed on the transduced CD34+ cells in the drug substance and on peripheral blood mononuclear cells (PBMC)
Adverse events | Up to 15 years post treatment
  Frequency and severity of clinical AEs and changes in laboratory parameters
Transgene copy number in the transduced CD34+ cells in the drug substance | At Day 0
  by qPCR
Change in total number of T cells | 6, 12, 24 months post treatment
  by flow cytometry
Change in distribution of different subpopulations | 6, 12, 24 months post treatment
  by flow cytometry, according to the WBC count: Naïve and activated/memory CD4+ and CD8+ T cells will be evaluated using CCR7/CD45RA/CD45RO markers. Early thymic emigrants will be monitored by detecting CD31+CD45RA+CD4+ T lymphocytes; Stem cell-like memory CD8+ and CD4+ T cells will be quantified by counting CCR7+CD45RA+CD8+ T cells. Evaluation of the distribution of TCRαβ and TCRγδ T cells
Change in T lymphocyte in vitro proliferation in the presence of mitogens and antigens | 6, 12, 24 months post treatment
Change in repertoire of T lymphocytes | 12, 24 months post treatment
  via high-throughput sequencing of the TCR
Evaluation of the B lymphocyte compartment | 6 months post treatment
  analysis of the circulating B cell subpopulations by flow cytometry: total CD19+ cells, naive (CD19+IgD+CD27-), switched memory (CD19+IgD-CD27+), marginal zone (CD19+IgD+CD27+), transitional (CD19+IgD+CD27-CD24highCD38+), 21low (CD19+CD38-CD21low). Immunoglobulin levels (IgG, A, M and E) and specific antibody production after immunization (if applicable)
Evaluation of the B lymphocyte compartment | At 12 months post treatment
  analysis of the circulating B cell subpopulations by flow cytometry: total CD19+ cells, naive (CD19+IgD+CD27-), switched memory (CD19+IgD-CD27+), marginal zone (CD19+IgD+CD27+), transitional (CD19+IgD+CD27-CD24highCD38+), 21low (CD19+CD38-CD21low). Immunoglobulin levels (IgG, A, M and E) and specific antibody production after immunization (if applicable)
Evaluation of the B lymphocyte compartment | At 24 months post treatment
  analysis of the circulating B cell subpopulations by flow cytometry: total CD19+ cells, naive (CD19+IgD+CD27-), switched memory (CD19+IgD-CD27+), marginal zone (CD19+IgD+CD27+), transitional (CD19+IgD+CD27-CD24highCD38+), 21low (CD19+CD38-CD21low). Immunoglobulin levels (IgG, A, M and E) and specific antibody production after immunization (if applicable)

SECONDARY OUTCOMES:
End of ongoing infection before the transplantation | Up to 15 years post treatment
Kinetics of immune reconstitution | Up to 15 years post treatment
  Kinetics of immune reconstitution
Adverse event | Up to 15 years post treatment
  Adverse event will be measured using CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra MAGNANI, MD, PhD, Study Director — Department of Biotherapy,LTCG, Necker-Enfants Malades Hospital; Chantal Lagresle-Peyrou, MD, Study Director — IMAGINE
Locations (1):
- Department of Pediatric Immunology, Hematology and Rheumatology UIHR, Necker-Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No